CLINICAL TRIAL: NCT05881993
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of CBP-4888 in Healthy, Non-Pregnant Female Subjects
Brief Title: Study of CBP-4888 in Healthy, Non-Pregnant Female Subjects
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Comanche Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBP-4888-100
Record Dates: First submitted 2023-05-09; First posted 2023-05-31 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteer Study

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBP-4888 (Experimental): CBP-4888 administered once as a subcutaneous dose.
  Interventions: Drug: CBP-4888
- Placebo (Placebo Comparator): Normal Saline administered once as a subcutaneous dose.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CBP-4888 — siRNA therapeutic
  Arms: CBP-4888
Other: Placebo — Normal Saline
  Arms: Placebo

SUMMARY:
This is a Phase I, first-in-human, single-center, randomized, double-blind, placebo-controlled, single ascending dose study to evaluate the safety, tolerability, and PK of ascending doses of CBP-4888.

DETAILED DESCRIPTION:
This study will involve female subjects meeting all inclusion criteria and no exclusion criteria. Cohorts of CBP-4888 are planned to be investigated in a sequential dose-escalation manner. Each cohort of subjects will be randomized to CBP-4888 to placebo and administered a single subcutaneous dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy non-pregnant female subjects
* Body mass index (BMI) ≥ 18.5 and ≤ 35.0 kg/m2
* Medically healthy, defined as having no clinically significant abnormal screening results including clinical laboratory evaluations, medical history, vital signs, ECG, and physical examination as deemed by the Investigator.

Exclusion Criteria:

* Screening blood pressure < 100/60 mmHg or > 140/90 mmHg
* Screening heart rate that is < 40 bpm or > 99 bpm
* Clinically significant ECG abnormality at screening
* Used prescription medication within 14 days prior to dosing
* Used over the counter (OTC) medications (including herbal products, nutritional supplements, dietary supplements, and/or vitamins) within 7 days prior to dosing
* Donated blood or had significant blood loss within 56 days prior to dosing

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — females
Enrollment: 45 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 30 days
  Number of participants with treatment-related adverse events
Pain at Site of Injection | 30 days
  Assessment of Pain on a 5 point scale (none, mild, moderate, severe or potentially life threatening)
Tenderness at Site of Injection | 30 Days
  Assessment of Tenderness on a 5 point scale (none, mild, moderate, severe or potentially life threatening)
Erythema at Site of Injection | 30 days
  Assessment of Erythema on a 5 point scale (none, mild, moderate, severe or potentially life threatening)
Swelling at Site of Injection | 30 Days
  Assessment of Swelling on a 5 point scale (none, mild, moderate, severe or potentially life threatening)

SECONDARY OUTCOMES:
Cmax of CBP-4888 | 30 days
  Peak Plasma Concentration
AUC of CBP-4888 | 30 days
  Area Under the Plasma Concentration Versus Time Curve
Tmax of CBP-4888 | 30 days
  Time to maximum plasma concentration

OTHER OUTCOMES:
Pharmacodynamics | 30 days
  Concentraion of sFLt-1

CONTACTS AND LOCATIONS:
Overall Officials: Allison August, MD, Study Director — Chief Medical Officer
Locations (1):
- Comanche Biopharma Clinical Research Site #1, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No